CLINICAL TRIAL: NCT04758559
Title: Usability of myfood24 in Clinical Populations
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Dietary Assessment Ltd (Unknown)
Responsible Party: Principal Investigator, Janet Cade, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 266347
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Gastroenterology Surgery; Colorectal Surgery; Weight Loss; Weight Change, Body
Keywords: diet monitoring; diet optimisation; nutrition
MeSH Terms: conditions — Weight Loss; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: Randomised into:
  Usual care; myfood24; myfood24 with automated suggestions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Placebo Comparator): Patients receive usual care concerning dietary advice.
  Interventions: Other: usual care
- myfood24 (Experimental): Patients receive myfood24 a new online app to support tracking of food and nutrient intakes, and allows patients and healthcare professionals to communicate, seeing results of intakes to promote healthy dietary behaviour changes.
  Interventions: Other: myfood24
- myfood24 + diet optimisation (Experimental): Personalised feedback. Patients use myfood24 with an additional feature of new technology providing guidance of how to optimise their diets against targets, using information they provide about current intakes.
  Interventions: Other: myfood24

INTERVENTIONS:
Other: myfood24 — An app to support monitoring of food and nutrient intake using robust validated methodology.
  Other Names: myfood24 + diet optimisation
  Arms: myfood24; myfood24 + diet optimisation
Other: usual care — Patients will receive standard advice as provided by the clinical team, this may or may not include nutrition.
  Arms: Usual care

SUMMARY:
Many patients would benefit from dietary/nutritional support to better manage their conditions but evaluating current intake in relation to personal targets is labour-intensive and often does not feature as part of clinical consultations.

Primary objective: test usability and acceptability of 'myfood24 Health' for monitoring dietary intake in a group of patients.

Recruit 60 gastroenterology surgery patient (Leeds) and 60 Tier 3 Weight Management patients (30 Leeds/ 30 York).

Randomise to 3 groups

1. usual care
2. myfood24Health
3. myfood24Health plus personalised feedback 'diet optimisation engine' which suggests changes to amounts or types of foods

During a 2-month follow-up, patients in group 2 or 3 will be asked to record daily diet in myfood24, including weekend and weekdays and use it a minimum of 4 times.

HCPs will be able to review diet/nutrients for group 2 and 3 patients and can support dietary change or nutritional goals, as part of patients' ongoing clinical management, during existing scheduled clinic visits (N.B. not all participants will have a scheduled clinic appointment during the study).

2 months after recruitment, all participants will receive a link to an online feedback questionnaire.

At end of study, HPCs will be invited to provide feedback during a 30 minute interview.

DETAILED DESCRIPTION:
See published results at https://www.mdpi.com/2072-6643/14/9/1768

ELIGIBILITY:
Inclusion Criteria:

* Able to use a smartphone or tablet
* Have regular access to the internet
* Aged 18 years or over
* Not receiving palliative treatment for their condition
* No pre-existing condition, eg. diabetes which requires a specific diet or eating disorder
* No food allergies
* Be receiving ongoing gastrointestinal surgery or weight management treatment
* Be able to read and understand English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Usability of myfood24 | 6 weeks
  System usability scale 1 to 10. HIgher score is better. Online survey.

SECONDARY OUTCOMES:
Ability of myfood24+ diet optimisation to change diet to meet diet targets | 6 weeks
  myfood24 app allows the healthcare professional to set personalised nutrition targets for the patient. Nutrient intakes will be measured in myfood24 and myfood24+ diet optimisation groups. We will explore differences in nutrient intakes between the groups. Nutrients measured will be daily intake average for energy (kcal), protein (g), fat (g), carbohydrate (g), fibre (g) sodium (g).
Response rate | 6 weeks
  response rates prior to undertaking a full scale randomised controlled trial
Correlation between diet and routine measure of body mass index | 6 weeks
  To explore correlations between mean energy intake (kcal/day) as recorded by multiple online 24-hour dietary recalls, with routine BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Gastroenterology surgery, Leeds, W. Yorks
  - Tier 3 Weight Management Clinic, York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wark PA, Hardie LJ, Frost GS, Alwan NA, Carter M, Elliott P, Ford HE, Hancock N, Morris MA, Mulla UZ, Noorwali EA, Petropoulou K, Murphy D, Potter GDM, Riboli E, Greenwood DC, Cade JE. Validity of an online 24-h recall tool (myfood24) for dietary assessment in population studies: comparison with biomarkers and standard interviews. BMC Med. 2018 Aug 9;16(1):136. doi: 10.1186/s12916-018-1113-8. PMID 30089491
- [Result] Carter MC, Albar SA, Morris MA, Mulla UZ, Hancock N, Evans CE, Alwan NA, Greenwood DC, Hardie LJ, Frost GS, Wark PA, Cade JE; myfood24 Consortium. Development of a UK Online 24-h Dietary Assessment Tool: myfood24. Nutrients. 2015 May 27;7(6):4016-32. doi: 10.3390/nu7064016. PMID 26024292
- See also: website of myfood24 tool — http://www.myfood24.org/